CLINICAL TRIAL: NCT07088302
Title: Effect OF Lactase Enzyme Supplements ON Protection Against Feeding Intolerance IN Preterm Neonates
Brief Title: Effect OF Lactase Enzyme Supplements ON Intolerance IN Preterm Neonates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Assistant professor of Pediatrics, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0108387
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Premature; Feeding Disorders; Lactase Deficiency, Congenital
MeSH Terms: conditions — Premature Birth; Feeding and Eating Disorders; Lactase Deficiency, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactase enzyme group (Active Comparator)
  Interventions: Drug: lactase administration
- Control group (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: lactase administration — 1 drop for each 10 ml of formula milk for 14 days
  Arms: Lactase enzyme group
Other: placebo — 10 ml milk without lactase
  Arms: Control group

SUMMARY:
This study aims to study the effect of lactase enzyme in preventing feeding intolerance in preterm neonates in neonatal intensive care unit at Alexandria University Children's Hospital.

ELIGIBILITY:
Inclusion criteria will be as follows:

* Preterm neonates ≤ 32 weeks gestational age.
* Start feeding in the first 72 hours of life. 8. Exclusion criteria

Patients with any of the following will be excluded:

1. Parental consent lacking/refusal.
2. Obvious major congenital abnormalities.
3. Infants more than 72 hours of age at the time of randomization.
4. Delayed introduction of feeding (beyond three days of life).
5. Known galactosemia.
6. Severe IUGR. -

Ages: 3 Days to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Feeding intolerance: | first two weeks of life
  vomiting number per day aspirates in ml/day abdominal distension by measuring abdominal circumference before and after feeds

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa Mohamed Farag, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided